CLINICAL TRIAL: NCT06753799
Title: The Effect of Education Based on Social Cognitive Learning Theory on Patient Participation, Self-Efficacy and Wound Healing in Individuals With Diabetic Foot Ulcer
Brief Title: The Effect of Education on Patient Care Outcomes in Individuals With Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fadime Koyuncu (Other)
Responsible Party: Sponsor-Investigator, Fadime Koyuncu, Principal Investigator, Research Assistant, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Organization: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SBUniversitesi2024
Record Dates: First submitted 2024-12-11; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Foot Ulcer, Diabetic; Patient Engagement; Self Efficacy; Wound Healing; Nursing
Keywords: Diabetic foot ulcer; patient participation; self-efficacy; wound healing; nursing
MeSH Terms: conditions — Diabetic Foot; Patient Participation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Active Comparator): The intervention group received training based on Social Cognitive Learning Theory
  Interventions: Behavioral: The intervention group received training based on Social Cognitive Learning Theory.
- The control group (No Intervention): The control group received routine clinical training (is in the form of verbal information)

INTERVENTIONS:
Behavioral: The intervention group received training based on Social Cognitive Learning Theory. — One of the theories that provides a conceptual framework for the learning and behavior change process is Social Cognitive Learning Theory. Verbal information is commonly provided in the education of individuals with diabetic foot ulcers. The difference of this study from other studies is that an educational booklet, an educational video and a demonstration method with a diabetic foot model are used during the education within the scope of theory-based education.
  Arms: The intervention group

SUMMARY:
The aim of this study is to determine the effect of Social Cognitive Learning Theory-based education on patient participation, self-efficacy and wound healing in individuals with diabetic foot ulcers. The research was conducted with 52 patients (25 intervention and 27 control) with Wagner 2 diabetic foot ulcers at Gülhane Training and Research Hospital between January and September 2024.

DETAILED DESCRIPTION:
The study was conducted in four stages: first application to the clinic, 1st month, 2nd month and 3rd month. While the Social Cognitive Learning Theory was applied to the intervention group, only the currrent clinical education was provided to the control group. The research data were collected using the "Data Collection Form Regarding Participants' Identifying Characteristics", "Diabetic Foot Information Form", "Metabolic Status and Wound Follow-up Form", "Patient Participation Scale" and "Diabetic Foot Care Self-Efficacy Scale". The results of this study show that education based on Social Cognitive Learning Theory is effective on patient participation, self-efficacy and wound healing in individuals with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older Agree to participate in the study Have type 2 diabetes Have a Wagner classification score of 2 Have the same wound care protocols (epidermal growth factor/hyalunoric acid containing cream and dressing with gauze)

Exclusion Criteria:

* Having communication difficulties and mental retardation Having vision and manual dexterity problems Having diabetic foot infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Change in ulcer size | From enrollment to the end of treatment at 3 months
  The result obtained by multiplying the length and width measurements of the ulcer with each other expresses the ulcer size in cm2.
Change in patient participation | From enrollment to the end of treatment at 3 months
  It was assessed with the Patient Health Engagement Scale (PHE-s). The PHE-s was developed based on a 4-stage model of patient. Items of the PHE-s: blackout, arousal, adhesion and eudaimonic project. Patients were asked to respond by positioning themselves between one and seven points in relation to their experience.
Change in self-efficacy | From enrollment to the end of treatment at 3 months
  "Participants achieved a response if they scored a self efficacy status of 0 or 10 on a scale ranging from 0 (worst outcome) to 90 (best outcome)."

CONTACTS AND LOCATIONS:
Overall Officials: Fadime Koyuncu, 2, Study Chair — University of Health Sciences Gulhane Faculty of Nursing; Kerim Bora YILMAZ, 3, Study Chair — Gulhane Training and Research Hospital
Locations (1):
- University of Health Sciences Gulhane Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
all collected IPD